CLINICAL TRIAL: NCT01612546
Title: Pilot Trial of CRLX101 in the Treatment of Patients With Advanced Gastric, Gastroesophageal, or Esophageal Squamous or Adenocarcinoma
Brief Title: Pilot Trial of CRLX101 in Treatment of Patients With Advanced or Metastatic Stomach, Gastroesophageal, or Esophageal Cancer That Cannot be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11276; NCI-2012-00893 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-06-04; First posted 2012-06-06 (Estimated); Results first posted 2017-12-27 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Adenocarcinoma of the Esophagus; Adenocarcinoma of the Gastroesophageal Junction; Diffuse Adenocarcinoma of the Stomach; Intestinal Adenocarcinoma of the Stomach; Mixed Adenocarcinoma of the Stomach; Recurrent Esophageal Cancer; Recurrent Gastric Cancer; Squamous Cell Carcinoma of the Esophagus; Stage IIIB Esophageal Cancer; Stage IIIB Gastric Cancer; Stage IIIC Esophageal Cancer; Stage IIIC Gastric Cancer; Stage IV Esophageal Cancer; Stage IV Gastric Cancer
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Esophageal Neoplasms; Stomach Neoplasms; Esophageal Squamous Cell Carcinoma | interventions — IT-101

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (cyclodextrin-based polymer-camptothecin CRLX101) (Experimental): Patients receive cyclodextrin-based polymer-camptothecin CRLX101 IV over 60 minutes on days 1 and 15. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity. After the completion of 6 courses, patients achieving stable disease or better may receive treatment for an additional 6 months.
  Interventions: Drug: cyclodextrin-based polymer-camptothecin CRLX101; Other: Laboratory biomarker analysis; Other: Pharmacological studies

INTERVENTIONS:
Drug: cyclodextrin-based polymer-camptothecin CRLX101 — Given IV
  Other Names: CRLX101; cyclodextrin-based polymer-camptothecin IT-101; IT-101
Other: Laboratory biomarker analysis — Correlative studies
Other: Pharmacological studies — Correlative studies

SUMMARY:
This pilot clinical trial studies cyclodextrin-based nanopharmaceutical CRLX101 in treating patients with advanced or metastatic stomach, gastroesophageal, or esophageal cancer that has progressed through at least one prior regimen of chemotherapy and cannot be removed by surgery. CRLX101 delivers the cytotoxic topoisomerase-1 inhibitor camptothecin into tumor cells and is hypothesized to interrupt the growth of tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate pre- and post-treatment biopsies to assess CRLX101 (cyclodextrin-based polymer-camptothecin CRLX101) nanoparticle and 20(S)-Camptothecin (CPT) uptake in tumor and normal tissue.

SECONDARY OBJECTIVES:

I. To evaluate the safety and toxicity of CRLX101 in this patient population.

II. To examine the antitumor efficacy of CRLX101 in advanced gastric/gastroesophageal junction (GEJ)/esophageal squamous or adenocarcinoma including clinical benefit rate (complete response [CR] + partial response [PR] + stable disease [SD]) at 4 months and overall survival.

OUTLINE:

Patients receive cyclodextrin-based polymer-camptothecin CRLX101 intravenously (IV) over 60 minutes on days 1 and 15. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.

Patients achieving stable disease or better, may receive treatment for an additional 6 months.

After completion of study treatment, patients are followed up monthly.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed advanced or metastatic squamous adenocarcinoma of the esophagus, GEJ, or stomach
* Patients must have primary tumor and adjacent normal tissue accessible via endoscopic biopsy
* Patients must have received at least one prior chemotherapy regimen for their unresectable or metastatic disease, not including treatment administered in the adjuvant and/or neoadjuvant setting for curative intent
* Patients must have measurable or evaluable disease
* Absolute neutrophil count >= 1500 cells/uL
* Platelets >= 100,000 cells/uL
* Total bilirubin =< 1.5 times the upper limit of normal (ULN)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x ULN
* AST/ALT =< 5 x ULN if liver metastasis is present
* Serum creatinine =< 1.5 mg/dL or a measured creatinine clearance >= 50 mL/min
* Prothrombin time (PT)/partial thromboplastin time (PTT) =< 1.5 x ULN
* Subjects with an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Subjects with a life expectancy >= 12 weeks
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately and be discontinued on study; subjects should be instructed to notify the investigator if it is determined after completion of the study that they became pregnant during the treatment phase of the study; the anticipated date or birth or termination of the pregnancy should be provided at the time of the initial report; whenever possible, a pregnancy should be followed to term, any premature terminations reported, and the status of the mother and the child should be reported to the study monitor after delivery; if the outcome of the pregnancy meets any severe adverse events (SAE) classification criterion, the investigator must follow the procedures for reporting SAEs; any neonatal death occurring =< 30 days after birth must also be reported as a SAE
* Subjects must have an electrocardiogram without evidence of clinically significant conduction abnormalities or active ischemia as determined by the investigator and an acceptable QTc interval
* All subjects must have the ability to understand and the willingness to sign a written informed consent
* Subjects must not have received prior chemotherapy or radiation within < 4 weeks prior to first dose of study drug
* Subjects may be entered if they have received prior radiation therapy involving =< 30% of the bone marrow; any prior radiation therapy must have been administered >= 4 weeks prior to first dose of study drug and the subject must be recovered from the acute toxic effects of the treatment prior to first dose of study drug (defined as a return to baseline or a severity of =< grade 1)
* Subjects may be enrolled with a history of treated brain metastases that are clinically stable for >= 4 weeks prior to the first dose of study drug; subjects may not be currently receiving dexamethasone

Exclusion Criteria:

* Female subjects who are pregnant or nursing
* Subjects who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to first dose of study drug or those who have not had adverse events return to baseline severity level or a severity of grade 1 due to agents administered more than 4 weeks prior to first dose of study drug
* Subjects with a history of congestive heart failure (CHF) requiring medical therapy
* Subjects with serum amylase or lipase > 1.5 ULN
* Subjects with previous high dose chemotherapy with autologous stem cell rescue bone marrow transplantation
* History of organ or allogeneic bone marrow transplant
* Use of any investigational agent or device within 4 weeks prior to first dose of study drug
* Metastatic disease to the central nervous system (CNS) requiring treatment or radiation therapy
* Subjects with known untreated brain metastases or treated brain metastases that have not been stable >= 4 weeks prior to first dose of study drug
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection (including human immunodeficiency virus [HIV] not stable on antiretroviral therapy), symptomatic congestive heart failure, hypertension, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements, as determined by the investigator
* History of prior malignancy not cured by excision; patients with non-melanoma skin cancer or carcinoma in situ of the cervix are not excluded, but patients with other prior malignancies must have had at least 2-year disease free interval
* Concurrent therapeutic anticoagulation: PTT less than or equal to 1.5 x ULN or low dose aspirin and low-molecular weight heparin only are allowed; Coumadin will be allowed on a case by case basis if use is chronic and approved by the study medical monitors
* Any major surgery =< 4 week prior to first dose of study drug
* Concurrent use of filgrastim (G-CSF) or growth factors at the time of initiation of study drug
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to CRLX101 and camptothecins
* Subjects with marked baseline prolongation of QT/QTc interval (for females QTc interval >= 470 msec and for males QTc interval >= 450 msec)
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-11; Primary Completion 2015-01-15 (Actual); Study Completion 2015-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Chao, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Cyclodextrin-based Polymer-camptothecin CRLX101): Patients receive cyclodextrin-based polymer-camptothecin CRLX101 IV over 60 minutes on days 1 and 15 at 15 mg/m^2. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity. After the completion of 6 courses, patients achieving stable disease or better may receive treatment for an additional 6 months.
  cyclodextrin-based polymer-camptothecin CRLX101: Given IV
  Laboratory biomarker analysis: Correlative studies
  Pharmacological studies: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Cyclodextrin-based Polymer-camptothecin CRLX101)
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Cyclodextrin-based Polymer-camptothecin CRLX101)
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 64 [48 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: CRLX101 (CPT) Uptake in Tumor and Nearby Normal Tissue
Description: Using Fisher's Exact to determine statistical significance in detection of a CPT fluorescence signal posttreatment between tumor and adjacent normal tissue biopsy specimens.
Time Frame: Baseline and day 8
Population: One patient was not included in the analysis because no tumor tissue was identified in the biopsy samples both pre and post-CRLX101 treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Cyclodextrin-based Polymer-camptothecin CRLX101)
Number analyzed (Participants) | 9
Participants
  CPT signal was observed in the tissue: Tumor tissue | 9
  CPT signal was observed in the tissue: Nonneoplastic tissue | 0
  CPT signal was not observed in the tissue: Tumor tissue | 0
  CPT signal was not observed in the tissue: Nonneoplastic tissue | 9
Statistical Analysis 1: Comparison: Treatment (Cyclodextrin-based Polymer-camptothecin CRLX101); Test type: Other; p < 0.01, Fisher Exact

2. Secondary Outcome: Overall Objective Response Rate
Description: Patients with best response of Complete Response or Partial Response assessed using Response Evaluation Criteria In Solid Tumors (RECIST) 1.1. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to 4 years
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Cyclodextrin-based Polymer-camptothecin CRLX101)
Number analyzed (Participants) | 10
percentage of participants | 0

3. Secondary Outcome: Clinical Benefit Rate
Description: Patients with a best response of Complete Response, Partial Response or Stable Disease after at least 4 months of treatment assessed using Response Evaluation Criteria In Solid Tumors (RECIST) 1.1. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), not a CR, PR, Progression or Symptomatic Deterioration; Progression (PD), a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; Symptomatic Deterioration, global deterioration of health status requiring discontinuation of treatment without objective evidence of progression. Clinical Benefit (CR + PR +SD≥4months).
Time Frame: At least 4 months post treatment, assessed up to 4 years
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Cyclodextrin-based Polymer-camptothecin CRLX101)
Number analyzed (Participants) | 10
percentage of participants | 10

4. Secondary Outcome: Overall Survival
Description: Estimated using the product-limit method of Kaplan and Meier.
Time Frame: From date of start of therapy to date of death due to any cause, assessed up to 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Cyclodextrin-based Polymer-camptothecin CRLX101)
Number analyzed (Participants) | 10
months | 5.5 [1.5 to 28.1]

5. Secondary Outcome: Incidence of Adverse Events
Description: Incidence of treatment related adverse events graded per NCI CTCAE version 4.03
Time Frame: Up to 4 years
Measure: Number; unit: participants
Arm/Group | Treatment (Cyclodextrin-based Polymer-camptothecin CRLX101)
Number analyzed (Participants) | 10
participants
  Grade 1 or 2 : Fatigue | 5
  Grade 1 or 2 : Nausea | 3
  Grade 1 or 2 : Proteinuria | 3
  Grade 1 or 2 : Hematuria | 2
  Grade 1 or 2 : Vomiting | 1
  Grade 1 or 2 : Diarrhea | 1
  Grade 1 or 2 : Infusion reaction | 1
  Grade 1 or 2 : Pruritus | 1
  Grade 1 or 2 : Myalgia | 1
  Grade 1 or 2 : Cystitis | 1
  Grade 1 or 2 : Cough | 1
  Grade 1 or 2 : Hypertension | 1
  Grade 1 or 2 : Alk Phos elevation | 1
  Grade 1 or 2 : AST elevation | 1
  Grade 1 or 2 : Cardiac chest pain | 0
  Grade 1 or 2 : Anemia | 3
  Grade 1 or 2 : Leukopenia | 2
  Grade 1 or 2 : Neutropenia | 2
  Grade 1 or 2 : Lymphopenia | 1
  Grade 1 or 2 : Thrombocytopenia | 1
  Grade 3 : Fatigue | 0
  Grade 3 : Nausea | 0
  Grade 3 : Proteinuria | 0
  Grade 3 : Hematuria | 0
  Grade 3 : Vomiting | 0
  Grade 3 : Diarrhea | 0
  Grade 3 : Infusion reaction | 0
  Grade 3 : Pruritus | 0
  Grade 3 : Myalgia | 0
  Grade 3 : Cystitis | 0
  Grade 3 : Cough | 0
  Grade 3 : Hypertension | 0
  Grade 3 : Alk Phos elevation | 0
  Grade 3 : AST elevation | 0
  Grade 3 : Cardiac chest pain | 1
  Grade 3 : Anemia | 0
  Grade 3 : Leukopenia | 0
  Grade 3 : Neutropenia | 0
  Grade 3 : Lymphopenia | 0
  Grade 3 : Thrombocytopenia | 0

ADVERSE EVENTS:
Time Frame: Adverse events collected over a period of 2 years.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Treatment (Cyclodextrin-based Polymer-camptothecin CRLX101)
Serious Adverse Events (participants affected / at risk) | 2/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Cyclodextrin-based Polymer-camptothecin CRLX101) (N=10)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Cyclodextrin-based Polymer-camptothecin CRLX101) (N=10)
Anemia (Blood and lymphatic system disorders) | 9 (18)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (3)
Sinus tachycardia (Cardiac disorders) | 5 (6)
Abdominal distension (Gastrointestinal disorders) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 5 (6)
Ascites (Gastrointestinal disorders) | 1 (2)
Bloating (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 4 (5)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (8)
Obstruction gastric (Gastrointestinal disorders) | 1 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (7)
hepatomegaly (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Edema limbs (General disorders) | 3 (4)
Fatigue (General disorders) | 8 (15)
Infusion related reaction (General disorders) | 1 (2)
Allergic reaction (Immune system disorders) | 1 (1)
Nail infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Activated partial thromboplastin time pr (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 5 (7)
Aspartate aminotransferase increased (Investigations) | 5 (8)
Lymphocyte count decreased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (10)
Platelet count decreased (Investigations) | 2 (2)
Weight loss (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 2 (8)
Alkalosis (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (7)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 5 (6)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 4 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (6)
Restless Leg Syndrome (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (3)
Hematuria (Renal and urinary disorders) | 2 (5)
Proteinuria (Renal and urinary disorders) | 4 (8)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
pale (Skin and subcutaneous tissue disorders) | 1 (1)
sweat (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 6 (18)
Hypotension (Vascular disorders) | 4 (5)
Thromboembolic event (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes